CLINICAL TRIAL: NCT05325580
Title: Intravenous Magnesium Sulfate Vs Placebo to Treat Non-traumatic Acute Headaches in the Emergency Department
Brief Title: Intravenous Magnesium Sulfate Vs Placebo to Treat Non -Traumatic Acute Headaches in the Emergency Department
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Pr.Semir Nouira chef of emergency deparment, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Emergency Monastir
Record Dates: First submitted 2022-03-16; First posted 2022-04-13 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-02

CONDITIONS: Head Pain
Keywords: intavenous; magnesium sulfate; nontraumatic; acute headaches; placebo
MeSH Terms: conditions — Headache | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): 1g paracetamol + 20 min infusion of 150ml of saline serum
  Interventions: Drug: Magnesium sulfate
- magnesium group (Experimental): 1g paracetamol + 20 min infusion of 2g magnesium in 150 ml of serum saline
  Interventions: Drug: Magnesium sulfate

INTERVENTIONS:
Drug: Magnesium sulfate — magnesium group 1g paracetamol + 20 min infusion of 2 g magnesium in 150 ml of saline serum and Placebo Group
  1g paracetamol + 20 min infusion of 150 ml of saline serum
  Other Names: placebo

SUMMARY:
Intravenous Magnesium Sulfate Vs Placebo to Treat Non -Traumatic Acute Headaches in the Emergency Department

DETAILED DESCRIPTION:
Rate of Intravenous Magnesium Sulfate Vs Placebo to Treat Non -Traumatic Acute Headaches in the Emergency Department

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* age >18 years
* Acute non-traumatic acute headaches
* patients treated in ED
* Magnesium sulfate and aspirin administered intravenously (IV)

Exclusion Criteria:

* Current regular use of analgesics, anticonvulsants or antidepressants
* Renal disorder with a low glomerular filtration rate (<60 ml/min)
* Neuromuscular disorder
* Pregnant woman
* Contrindication
* Allergy to NSAID
* Traumatic Headache
* Chronic headache ( headache occurring at least 15 days per month for at least 3 months)
* Hemodynamic instability

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Intravenous Magnesium Sulfate to Treat Non -Traumatic Acute Headaches in the Emergency Department | 1day
  Patients with Non -Traumatic Acute Headaches in the Emergency Department recived 1g paracetamol + 20 min infusion of 2g magnesium

SECONDARY OUTCOMES:
Placebo to Treat Non -Traumatic Acute Headaches in the Emergency Department | 1 day
  Patients with Non -Traumatic Acute Headaches in the Emergency Department received 1g paracetamol + 20 min infusion of saline serum

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, Professor, Principal Investigator — University of Monastir
Locations (1):
- University of Monasrtir, Monastir, Tunisia